CLINICAL TRIAL: NCT05972525
Title: What Matters to Patients With Severe Hip or Knee Osteoarthritis? Decisional Quality, Patient Involvement and Health Outcome
Brief Title: What Matters to Patients With Severe Hip or Knee Osteoarthritis?
Acronym: PATI-Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S-20200137
Record Dates: First submitted 2023-06-08; First posted 2023-08-02 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Hip Osteoarthritis; Knee Osteoarthritis; Shared Decision Making; Total knee arthroplasty; Partiel knee arthroplasty; Total hip arthroplasty; Decision quality; HK-DQI
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The group of hip and knee surgeons at Vejle, Odense, and Svendborg hospitals will be randomized 1:1 either to continue standard consultation or to practice SDM supported by the in-consultation PtDA.
Who Masked: Outcomes Assessor
Masking Description: The external statistician will be blinded and responsible for performing the analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared decision-making (SDM) (Experimental): Patients will be informed by a nurse before being consulted by the surgeon randomized to SDM and use the in-consultation PtDA during the consultation on patients with severe hip or knee osteoarthritis
  Interventions: Behavioral: Shared decision-making supported by an in-consultation PtDA to patients with severe osteoarthritis in their hip or knee
- Usual practice (No Intervention): Patients will be informed by a nurse before being consulted by the surgeon randomized to usual practice during the consultation on patients with severe hip or knee osteoarthritis

INTERVENTIONS:
Behavioral: Shared decision-making supported by an in-consultation PtDA to patients with severe osteoarthritis in their hip or knee — The intervention group has been involved in the development process of the PtDA. After receiving a training course in SDM and the use of a PtDA, the surgeons will practice SDM supported by an in-consultation PtDA during the consultations with the participant.
  Arms: Shared decision-making (SDM)

SUMMARY:
This clinical trial aims to investigate if shared decision-making, and the use of an in-consultation patient decision aid (PtDA), increases the decisional quality and therefore treatment satisfaction and outcome of patients with severe hip or knee osteoarthritis.

Finally, an evaluation will be conducted on patient-reported outcomes on pain, physical function, quality of life (QoL), and patient satisfaction, up to one year after surgery.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common joint disease and a major cause of disability worldwide. The condition typically affects the hip or knee, and as the condition progresses it frequently causes debilitating pain and stiffness in the affected joints; thus impairing mobility, and decreasing function and quality of life(QoL).

Approximately 10,300 primary hip arthroplasties (THA) and 10,000 primary knee arthroplasties (TKA/UKA) were performed in Denmark in 2021.

For the majority of patients with severe osteoarthritis, evidence shows that joint replacement surgery is life-changing. Despite this documented effect, not all patients achieve optimal results. Patient dissatisfaction following THA and TKA has been reported as 7 % and 11-18%, respectively.

It is hypothesized that a lack of adequate information and patient involvement in the decision process might lead to the misalignment of patients' expectations and subsequent dissatisfaction. Considerable evidence shows that patients prefer more information and greater involvement. This strongly supports the concept that patients need to be actively involved in treatment decisions.

Accordingly, increasing patient involvement in healthcare decisions may be beneficial. Shared decision-making (SDM) supports patients' active involvement in the process and improves the quality of decisions. SDM can be facilitated using a PtDA, which has shown significant benefits in a range of patient groups. However, research on SDM and PtDAs in patients with severe hip or knee OA is lacking.

The overall aim of this project is to investigate if an in-consultation PtDA increases the decision quality for patients with severe OA of the hip or knee.

ELIGIBILITY:
Inclusion Criteria:

* Severe primary osteoarthritis eligible for primary total hip arthroplasty (THA) / primary total knee arthroplasty (TKA) / primary partial knee arthroplasty (UKA)
* Able to understand and read Danish
* Informed consent

Exclusion Criteria:

* Previous THA, TKA, or UKA on the contralateral side
* Cognitive impairment
* Non-OA-related reason for the visit
* No digital mailbox (E-boks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
The participant's decisional quality according to The Hip/Knee Osteoarthritis Decision Quality Instrument (HK-DQI). | Within one week after inclusion in the consultation
  Informed Patient-Centered (IPC) decision is calculated as the percentage of patients who are well-informed and received their preferred treatment.

SECONDARY OUTCOMES:
Participant's engagement in the decision-making process as measured by the CollaboRATE questionnaire | Within one week after inclusion in the consultation
  Minimum value: 0. Maximum value: 100. The higher the value the more shared decision-making
Participant's involvement in the decision-making process as measured by the HK-DQI questionnaire | Within one week after inclusion in the consultation
  HK-DQI, section 3, decision-making process: Minimum value: 0. Maximum value: 100. The higher the value the more shared decision-making
The duration of consultation when PtDA is used compared to standard consultation without the use of PtDA. | Through study completion, an average of 1 year
  The time duration will be documented by the surgeons

OTHER OUTCOMES:
Participant's Qol when undergoing hip or knee replacement surgery as measured by EuroQol (EQ-5D) | Three months and one year following surgery.
  QoL: EuroQol (EQ-5D): Measuring the health-related quality of life. Presenting in three levels; Level 1: Indicating no problem, to Level 3: Indicating extreme problems
The participant's pain and physical function after undergoing hip replacement surgery as measured by the Oxford Hip Score (OHS) questionnaire | Three months and one year following surgery
  Oxford Hip Score (OHS): Measuring function and pain with patients undergoing hip replacement surgery. Total scores range from 0 (poorest function) to 48 (maximal function).
The participant's pain and physical function after undergoing knee replacement surgery as measured by the Oxford Knee Score (OKS) questionnaire | Three months and one year following surgery
  Oxford Knee Score (OKS): Measuring function and pain with patients undergoing knee replacement surgery. Total scores range from 0 (poorest function) to 48 (maximal function).
The participant's physical function after undergoing hip or knee replacement surgery as measured by Forgotten Joint Score (FJS) questionnaire | Three months and one year following surgery.
  Forgotten joint score (FJS): Measuring the participants' awareness of their artificial joint during activity of daily living (ADL). Minimum value: 0. Maximum value: 100. The higher score, the less the patient is aware of their affected joint.
Participant's regret of the treatment decision as measured by the Decision Regret Scale questionnaire. | Three months and one year following surgery.
  The Decision Regret Scale: Minimum value: 0. Maximum value: 100. The higher the value the more regret.
Participant's satisfaction after undergoing hip or knee replacement surgery as measured by the patient satisfaction questionnaire (PSQ) | Three months and one year following surgery.
  The patient satisfaction questionnaire (PSQ): The higher the value the more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Ahlmann, PhD stud, Principal Investigator — Vejle Hospital; Claus Varnum, Ass.Prof.MD, Study Chair — Vejle Hospital; Martin Lindberg-Larsen, Ass.Prof.MD., Study Chair — Odense University Hospital; Charlotte Myhre Jensen, Ass.Prof.RN, Study Chair — Odense University Hospital; Karina Dahl Steffensen, Prof.MD., Study Chair — Vejle Hospital
Locations (3):
- Denmark (3):
  - Odense University Hospital, OUH, Odense
  - Odense University Hospital, OUH, Svendborg
  - Lillebaelt Hospital - Vejle, Vejle

IPD SHARING:
Plan to Share IPD: Yes
All data of the outcome measures will be available in an anonymized form if required by the scientific journal, in which the results of the trial will be published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after the publication of the trial
Access Criteria: Data access will be reviewed by the author's group

REFERENCES:
- [Derived] Pedersen TA, Lindberg-Larsen M, Jensen CM, Timm S, Steffensen KD, Varnum C. Impact of an in-consult patient decision aid on decisional quality, involvement, and health outcome for patients with severe hip or knee osteoarthritis - a study protocol for a multicentre, cluster randomised controlled trial (PATI-study). BMC Musculoskelet Disord. 2025 Jul 2;26(1):584. doi: 10.1186/s12891-025-08856-w. PMID 40597226

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05972525/SAP_001.pdf